CLINICAL TRIAL: NCT00850005
Title: IVIG for Treatment of Resistant Neuropathic Pain: a Preliminary Study
Brief Title: Intravenous Immunoglobulin (IVIG) for Resistant Neuropathic Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Alexander J Clark MD FRCPC, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 200434
Record Dates: First submitted 2009-02-18; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; resistant; neuroinflammation; neuroinflammatory markers; Neuropathic pain that has not responded to standard therapy
MeSH Terms: conditions — Neuralgia; Neuroinflammatory Diseases | interventions — Immunoglobulins, Intravenous; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVIG (Experimental): Active treatment will be intravenous immunoglobulin G (Gamunex, immune globulin intravenous [human], 10%), at a dose of 2 g/kg divided over five days (0.4 g/kg/day).
  Interventions: Biological: Intravenous immunoglobulin
- Placebo (Placebo Comparator): The placebo treatment will be intravenous normal saline and will be infused in a similar manner.
  Interventions: Biological: Normal Saline

INTERVENTIONS:
Biological: Intravenous immunoglobulin — 2 g/kg divided over five days
  Arms: IVIG
Biological: Normal Saline — Same volume as experimental arm
  Arms: Placebo

SUMMARY:
This project addresses a vexing problem that has alluded the best efforts of the medical/scientific community: treatment of resistant neuropathic pain. Neuropathic pain is common and includes conditions such as diabetic neuropathy, post herpetic neuralgia and post stroke pain and is believed to affect at least 3% of adults. Surveys of patients with neuropathic pain indicate that 60% do not receive adequate relief with current treatment. Results from recent laboratory and human studies reveal a new approach to treatment. This approach is based on the findings that neuroinflammation appears to be involved in development and maintenance of neuropathic pain. This study explores the effects of an immune-modulating blood-derived product, intravenous immunoglobulin (IVIG), in treating neuropathic pain. IVIG is thought to reduce neuroinflammation contributing to neuropathic pain. If successful, the study will provide important insights into pain mechanisms and a better understanding of how IVIG relieves neuropathic pain.

Hypotheses:

1. Reduction in neuroinflammation (NI) markers will co-vary with clinical indicators of pain relief
2. Patients with higher levels of markers of NI will be more likely to respond to IVIG

DETAILED DESCRIPTION:
This study will employ a randomized double blind cross-over design. A total of 12 subjects will be recruited for the study. Once each subject has satisfied the inclusion and exclusion criteria and provided informed consent, the subject will be randomized to either the IVIG or placebo treatment groups, using a pre-determined randomization list generated by the research office at the University of Calgary. Complete responders will begin a monitoring phase, partial and non-responders will return for a second cycle in one month. Complete responders, with prolonged relief, will cross-over to the alternative treatment when their pain returns if this occurs within 6 months of the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years; Clinical diagnosis of treatment-resistant neuropathic pain;
* Score of 4/10 or greater on the DN4 NeP screening questionnaire;
* Bedside examination confirming symptoms of neuropathic pain;
* Moderate to severe pain;
* Completed adequate analgesic trials according to neuropathic pain clinical practice guidelines;
* provides informed consent

Exclusion Criteria:

* Pregnant or lactating women;
* Clinical diagnosis of phantom limb pain;
* History of psychosis;
* current, substance dependency disorder;
* presence of clinically significant cardiac or pulmonary disorder that would compromise participants' safety;
* severe pain disorder other than the chronic NeP under study;
* Abnormalities above 1.5 times upper range of normal on screening CBC, blood chemistry;
* Serum IgA less than <0.05 g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-07 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will consist of change in mean daily pain diary score from baseline to each week post-treatment | Performed at screening, before the initial infusion, 2 weeks and 4 weeks post treatment

SECONDARY OUTCOMES:
Measurement of neuroinflammation (NI) markers (IL-1β, IL-6, IL-8, TNF-α, MMP-9, TIMP-1) | Performed at screening, before the initial infusion, 2 weeks and 4 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Clark, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada